CLINICAL TRIAL: NCT04931251
Title: Addressing Cancer-Related Financial Toxicity in Rural North Carolina Oncology Care Settings
Brief Title: Addressing Cancer-Related Financial Toxicity in Rural Oncology Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC1941; 5R01CA240092 (NIH); P30CA016086 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Neoplasms; Carcinoma
Keywords: Financial Toxicity; Cancer; Financial Navigation; Carcinoma; Neoplasms
MeSH Terms: conditions — Neoplasms; Carcinoma; Financial Stress

STUDY DESIGN:
Intervention Model Description: This is a multi-site, single arm, financial navigation intervention
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Financial Navigation (Other): includes a financial toxicity screening measure (COST), baseline and post-intervention surveys, and approximately 2-6 visits with a financial navigator to identify financial assistance resources
  Interventions: Behavioral: Financial Navigation

INTERVENTIONS:
Behavioral: Financial Navigation — providing financial navigation for cancer patients in NC to identify available financial assistance resources to assist patients with the cost of cancer

SUMMARY:
The financial burden, or financial toxicity (FT), of cancer is a consequential and growing problem, particularly for rural patients. It is important to improve our understanding of how financial navigation (FN) can reduce the material, psychological, and behavioral burden of costs associated with cancer care in both rural and non-rural community settings. The purpose of this study is to conduct a financial navigation program in 5 rural and 4 non-rural oncology practices in North Carolina and evaluate the effects of financial navigation on patient outcomes, including financial toxicity and health-related quality of life.

DETAILED DESCRIPTION:
This study is designed to evaluate the implementation and effectiveness of a financial navigation intervention within 5 rural and 4 non-rural oncology settings in North Carolina. Financial navigators from each of the 9 sites will recruit and enroll 255 patients total across all sites into a financial navigation program. The financial navigation intervention consists of screening patients using the COST measure for financial toxicity. If the patient scores 23 or lower, they are considered to have moderate to severe financial toxicity and will be enrolled in the study. Patients will then complete a series of baseline questionnaires to measure their health related quality of life and then they will meet with a financial navigator for a comprehensive intake process to determine potential financial assistance resources the patient may be eligible for and continued visits with the financial navigator until all financial assistance resources have been explored and patients have received benefits or referrals to financial assistance programs. At the end of the intervention, the patients will complete the COST measure again, and repeat baseline surveys to measure health-related quality of life and the patient's acceptability and responsiveness of the financial navigation intervention. Patient participation depends on the depth of patient need but ranges from 2 visits to 6 visits with the financial navigator over approximately 4 months but possibly longer depending on the complexity of the patient's financial need.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Patients with any type of cancer diagnosed within 5 years and/or living with advanced disease
* Patients who score 22 or lower on the COST measure indicating high FT
* Patients must be able to read and speak English

Exclusion Criteria:

* Participants without a cancer diagnosis
* Patients diagnosed more than 5 years ago without advanced disease
* Patients or caregivers under the age of 18
* Patients who do not sign the consent form
* Patients who do not complete the baseline COST survey
* Patients who cannot read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
COST (Comprehensive Score for Financial Toxicity) measure | 4-6 months
  To evaluate the change from baseline to follow-up in scores from the Comprehensive Score for Financial Toxicity (COST) measure after participation in the financial navigation program among 780 rural and non-rural NC cancer patients with high baseline financial distress.

SECONDARY OUTCOMES:
Health-Related Quality of Life (HrQoL) Measures | 4-6 months
  To evaluate the change from baseline to follow-up in scores from HRQoL, care-altering behaviors and patient perspectives on the intervention itself

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Wheeler, PhD, Principal Investigator — Lineberger Comprehensive Cancer Center, University of North Carolina at Chapel Hill
Locations (8):
- United States (8):
  - NC Basnight Cancer Hospital, Chapel Hill, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Vidant Medical Center, Cancer Center, Greenville, North Carolina
  - Pardee UNC Health Care, Pardee Cancer Center, Hendersonville, North Carolina
  - UNC Lenoir Cancer Care Services, Kinston, North Carolina
  - Carteret Health Care Cancer Center, Morehead City, North Carolina
  - The Outer Banks Hospital, Nags Head, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
We commit to broadly sharing appropriate materials and de-identified data that are developed with support from the NIH, while protecting participant privacy and confidentiality in accordance with best human subjects research practices and Health Insurance Portability and Accountability Act (HIPAA) guidelines. We commit to the collection, cataloging, protecting, and sharing of clinical and other research data and resources that is consistent with NIH policies, using the Research Electronic Data Capture (REDCap) platform as the mechanism for data storage, protection and sharing. We will only share de-identified IPD.
Supporting Information: Study Protocol
Time Frame: The de-identified data will become available after study completion.
Access Criteria: The access criteria for accessing our de-identified participant data is still being developed.

REFERENCES:
- [Background] Wheeler SB, Biddell CB, Manning ML, Gellin MS, Padilla NR, Spees LP, Rogers CD, Rodriguez-O'Donnell J, Samuel-Ryals C, Birken SA, Reeder-Hayes KE, Petermann VM, Deal AM, Rosenstein DL. Lessening the Impact of Financial Toxicity (LIFT): a protocol for a multi-site, single-arm trial examining the effect of financial navigation on financial toxicity in adult patients with cancer in rural and non-rural settings. Trials. 2022 Oct 3;23(1):839. doi: 10.1186/s13063-022-06745-4. PMID 36192802
- [Background] Planey AM, Spees LP, Biddell CB, Waters A, Jones EP, Hecht HK, Rosenstein D, Wheeler SB. The intersection of travel burdens and financial hardship in cancer care: a scoping review. JNCI Cancer Spectr. 2024 Sep 2;8(5):pkae093. doi: 10.1093/jncics/pkae093. PMID 39361410
- [Background] Wheeler SB, Thom B, Waters AR, Shankaran V. Interventions to Address Cancer-Related Financial Hardship: A Scoping Review and Call to Action. JCO Oncol Pract. 2025 Jan;21(1):29-40. doi: 10.1200/OP.24.00375. Epub 2025 Jan 10. PMID 39793544
- [Background] Wheeler SB, Manning ML, Gellin M, Padilla N, Spees LP, Biddell CB, Petermann V, Deal A, Rogers C, Rodriguez-O'Donnell J, Samuel-Ryals C, Reeder-Hayes K, Rosenstein DL. Impact of a Comprehensive Financial Navigation Intervention to Reduce Cancer-Related Financial Toxicity. J Natl Compr Canc Netw. 2024 Oct;22(8):557-562. doi: 10.6004/jnccn.2024.7030. PMID 39413831
- [Result] Wheeler SB, Birken SA, Wagi CR, Manning ML, Gellin M, Padilla N, Rogers C, Rodriguez J, Biddell CB, Strom C, Bell RA, Rosenstein DL. Core functions of a financial navigation intervention: An in-depth assessment of the Lessening the Impact of Financial Toxicity (LIFT) intervention to inform adaptation and scale-up in diverse oncology care settings. Front Health Serv. 2022 Nov 9;2:958831. doi: 10.3389/frhs.2022.958831. eCollection 2022. PMID 36925862
- [Result] Petermann VM, Biddell CB, Planey AM, Spees LP, Rosenstein DL, Manning M, Gellin M, Padilla N, Samuel-Ryals CA, Birken SA, Reeder-Hayes K, Deal AM, Cabarrus K, Bell RA, Strom C, Young TH, King S, Leutner B, Vestal D, Wheeler SB. Assessing the pre-implementation context for financial navigation in rural and non-rural oncology clinics. Front Health Serv. 2023 Oct 23;3:1148887. doi: 10.3389/frhs.2023.1148887. eCollection 2023. PMID 37941608
- [Result] Biddell CB, Spees LP, Petermann V, Rosenstein DL, Manning M, Gellin M, Padilla N, Samuel-Ryals CA, Birken SA, Reeder-Hayes K, Deal AM, Cabarrus K, Bell RA, Strom C, DeAntonio PA, Young TH, King S, Leutner B, Vestal D, Wheeler SB. Financial Assistance Processes and Mechanisms in Rural and Nonrural Oncology Care Settings. JCO Oncol Pract. 2022 Sep;18(9):e1392-e1406. doi: 10.1200/OP.21.00894. Epub 2022 May 12. PMID 35549521
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials